CLINICAL TRIAL: NCT01155596
Title: Phase 2 Study of Negative Pressure Ventilation That Imapcts Weaning Ventilator in Medical Intensive Care Units
Brief Title: Negative Pressure Ventilation Imapcts Weaning Ventilator In Medical Intensive Care Units (ICUs)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Horng-Chyuan Lin/ Chief of Division of Pulmonary Infection and Immunity, Department of Thoracic Medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 98-3276B
Record Dates: First submitted 2010-05-30; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-06

CONDITIONS: Respiratory Failure
Keywords: Acute respiratory failure patients in medical ICUs.
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Base on positive pressure ventilation with intubation and mechanical ventilator, weaning processes will undergo by Pulmonologists.
- Experimental group (Experimental): Experimental group is weaning with the support of negative pressure ventilator.
  Interventions: Behavioral: negative pressure ventilator use

INTERVENTIONS:
Behavioral: negative pressure ventilator use — Body ventilators that assist ventilation by applying intermittent subatmospheric pressure around the thorax, abdomen, or airway and periodically expand the chest wall and inflate the lungs. They are relatively simple to operate and do not require tracheostomy. Chest cuirass is used in this study.
  Arms: Experimental group

SUMMARY:
This is a Quasi-experimental research design. The subjects are limited in intensive care unit within north medical center hospital. All subjects depend on ventilator and receive weaning plans. Experimental group is weaning with the support of negative pressure ventilator .The investigators collect basic personal variables in the questionnaire, APACHE Ⅱ scale, Dyspnea scale and arterial blood gas analysis and ventilator weaning index. Compare experimental group and control group data. Data will be Statistical analyzed by: descriptive statistics (such as: mean, standard deviation, median, frequency, percentage) and inferential statistics (such as: Independent T-test, Pair T-test, Mann-Whitney U test), P-value <0.05 will consider to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure patients in medical ICUs

Exclusion Criteria:

* Age<20 years old
* Malignancy
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Ventilator weaning rate | 28 days

SECONDARY OUTCOMES:
ICU stay | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Gung Memorial Hospital, Chang Gung University, College of Medicine., Taipei, Taiwan